CLINICAL TRIAL: NCT04236232
Title: The Impact of Subclinical Hypothyroidism on the Cardiovascular System
Brief Title: The Impact of Subclinical Hypothyroidism on Cardiovascular System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Randa Mahrous Roushdy, Resident doctor, Assiut University
Other Study IDs: Subclinical Hypothyroidism
Record Dates: First submitted 2019-09-24; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroid Function Tests; Ultrasonography, Carotid Arteries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who will be diagnosed as Subclinical Hypothyroidism: 50 pt who will be diagnosed as Subclinical Hypothyroidism by elevated level of TSH (TSH: >4.5 mu/l) and normal T4
  Interventions: Diagnostic Test: Thyroid function
- Patients with normal thyroid function: 50 pt with normal thyroid function (TSH &T4)
  Interventions: Diagnostic Test: Thyroid function

INTERVENTIONS:
Diagnostic Test: Thyroid function — Thyroid function,Lipid Profile, systolic Blood pressure ,diastolic blood pressure .Body Mass Index ,CRP,Echocardiography،ECG, Ultrasonography of Carotid artery
  Other Names: Thyroid function,Lipid Profile, systolic Blood pressure ,diastolic blood pressure .Body Mass Index ,CRP,Echocardiography،ECG, Ultrasonography of Carotid artery

SUMMARY:
This research aims to evaluate the relation between SCH and cardiovascular System by assessment of lipid profile and carotid intima-media thickness (CIMT), as a marker of atherosclerosis, and endothelial function.

DETAILED DESCRIPTION:
Subclinical hypothyroidism (SCH) is defined as a condition that characterized by elevated serum thyroid-stimulating hormone (TSH) concentrations (TSH: >4.5 mu/l), while circulating thyroxine (T4) and tri- iodothyronine (T3) levels remain within the normal range.

Depending on the extent of serum TSH elevation, SCH can be divided into Mild (where the concentration of serum TSH is in the range of 4.5-9 mU/l) Severe (TSH≥10 mU/l) SCH. Mild SCH constitutes ~75% of the total number of patients with SCH. The incidence of SCH varies between 5 and 10 % depending upon the gender, age, more frequent in women than in men, with increasing prevalence with advanced age in both sexes The consequences of SCH are variable at several levels and may depend on the duration and the degree of increasing level of the serum TSH. However, a number of important questions about SCH remain, including whether it increases cardiovascular (CVS) risk or not.

SCH has many causes the most common (60% to 80%) is chronic autoimmune thyroiditis associated with the presence of circulating anti-thyroid peroxidase antibodies(TPOAb) that are the most sensitive serological test for thyroid autoimmunity and/or antithyroglobulin Antibodies(TgAb).

The association between subclinical hypothyroidism (SCH) and cardiovascular disease has received increasing attention in recent years.

Thyroid hormones exert a direct effect on the heart and blood vessels. The deficit of these hormones leads to functional disorders of the Cardiovascular System (CVS) such as changes in cardiac frequency, cardiac output, left ventricular diastolic dysfunction, and reduced resting and exceptional systolic function.

Vascular abnormalities, such as increased vascular resistance, arterial stiffness, endothelial dysfunction, that is considered to be an early step in the development and progression of atherosclerosis.

The early changes in patients with SCH is alteration in lipid profile that could be a contributing factor for the risk of atherosclerosis, hyperlipidemia is one of the common causal factors of endothelial dysfunction.

Elevation of TSH has a positive correlation with serum total cholesterol (TC), triglycerides, LDL cholesterol (LDL-C), and a negative correlation to HDL cholesterol.

Some studies found significant lipid profile changes in patients with SCH, some others did not.

Atherosclerosis is a diffuse, degenerative disease of the arteries that results in the formation of porridge-like lipid deposit plaques in the great arterial wall, and accounts for the majority of cardiovascular disease incidence. Therefore, this association is the first to be assessed for the link between SCH and cardiovascular disease.

Progression of atherosclerosis features a chronic unresolved inflammatory response, leading to stenosis, embolization and thrombosis, since atherosclerosis is a chronic disease, to observe the whole pathogenesis in one single investigation would require a long time of study .Thus, endothelial dysfunction, as one of the earliest signs for atherosclerosis, could be most frequently observed in clinical investigation Assessment of endothelial dysfunction, being an early biomarker, is helpful in predicting cardiovascular risk by Carotid artery intima-media thickness (CIMT) measurement that has increasingly been used as a marker of atherosclerosis in many studies.

Evidence supporting the correlation between SCH and atherosclerosis has been accumulating:

The first study regarding the associated cardiovascular risk in patients with SCH was the long-time large cross-sectional Rotterdam study in the Netherlands, which showed an increased risk for atherosclerosis and prevalence of myocardial infarction among female patients with SCH aged >55 years. Velkoska and his colleagues who reported that SCH is associated with increase in CIMT and presence of carotid plaques independent of traditional atherosclerosis risk factors, Onder et al. who showed lack of a significant difference in CIMT between over and subclinical hypothyroid, indicating that the inflammation leading to increased CIMT starts in the subclinical phase .

ELIGIBILITY:
Inclusion Criteria:

* All healthy adult who will be diagnosed as SCH along with age ≥18 & gender-matched healthy relatives with normal thyroid function will be screened for evidence of high cardiovascular risk.

Exclusion Criteria:

* Hypo or hyper-thyroidism, Diabetes, Hypertension, cardiovascular disease, smokers, pregnant and lactating women.

Patients who had been treated with anti-thyroid drugs, radio iodine therapy or thyroxin hormone supplement or who had under gone thyroid surgery, those with a history of thyroid cancer or head and neck malignancies.

Those with history of drug use such as Contraceptive pill, Anti-depressant drugs, Corticosteroids, Anti arrhythmic drugs.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: patients who will be diagnosed as SCH, will present to Outpatient clinic of Assiut University hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Our data will reveale that SCH is associated with increase in CIMT and presence of carotid plaques,and these patients have an increased risk of cardiovascular disease compared with healthy patients. | Baseline
  The study Will include 50 patients with newly diagnosed SCH, and 50 healthy controls. Body mass index (BMI), TSH, fT4, lipids, blood pressure, mean and maximum carotid intima-media thickness (CIMT) will be determined in all participants.

REFERENCES:
- [Background] Sun J, Yao L, Fang Y, Yang R, Chen Y, Yang K, Tian L. Relationship between Subclinical Thyroid Dysfunction and the Risk of Cardiovascular Outcomes: A Systematic Review and Meta-Analysis of Prospective Cohort Studies. Int J Endocrinol. 2017;2017:8130796. doi: 10.1155/2017/8130796. Epub 2017 Aug 31. PMID 29081800
- [Background] Floriani C, Gencer B, Collet TH, Rodondi N. Subclinical thyroid dysfunction and cardiovascular diseases: 2016 update. Eur Heart J. 2018 Feb 14;39(7):503-507. doi: 10.1093/eurheartj/ehx050. PMID 28329380